CLINICAL TRIAL: NCT03495830
Title: Observational Multicentre Clinical Trial for Validation of Taxinomisis, New Stratification Tool for Stroke Risk in Patients With Carotid Disease
Brief Title: Stratification of Patient With Carotid Disease
Acronym: TAXINOMISIS
Status: Completed | Type: Observational
Sponsor: University of Belgrade (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); University of Barcelona (Other); University of Athens (Other); University of Genova (Other); Utrecht University (Other)
Responsible Party: Principal Investigator, Igor Koncar, Vascular surgeon,PhD, MD, University of Belgrade
Other Study IDs: STRATIFY; 755320 (Other Grant/Funding Number: European Union's Horizon 2020)
Record Dates: First submitted 2018-03-21; First posted 2018-04-12 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2022-01

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — At the inclusion in study, after 12,24 and 36 months blood samples will be analyzed, while 10 ml of blood sample will be stored for further analysis.
  Patients treated with carotid endarterectomy will have their plaque stored and analysed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Carotid endarterectomy: Patients that underwent intervention (CEA or CAS) are followed by clinical examination and carotid duplex on 12, 24 and 36 month If there is coexisting contralateral carotid stenosis with grade greater than 50% and not requiring interventional treatment (CEA or CAS), patient should cross in optimal medical therapy group.
  Interventions: Procedure: Carotid endarterectomy
- Optimal medical therapy group: Patients not subjected to intervention (or in whom one carotid has been treated with CAS or CEA and contralateral has stenosis is greater than 50%) will be followed with carotid duplex (at 12, 24 and 36 months) and MRI imaging of carotid tree from aortic arch up to the circle of Willis after 12 and 36 months.
  Interventions: Procedure: Carotid endarterectomy

INTERVENTIONS:
Procedure: Carotid endarterectomy — Exploration of carotid bifurcation. Clamping of carotid artery and plaque removal with endarterectomy. Plaque is stored. Suture of artery with direct suture or patch.

SUMMARY:
Introduction: Taxinomisis trial is part of the Taxinomisis project. The concept of the Taxinomisis project is to stratify carotid artery disease relying on new modern data corresponding to contemporary patients based on information from longitudinal studies. Taxinomisis trial will validate this tool and adjust such stratification. Initial step of the project is characterization of symptomatic and asymptomatic carotid atherosclerotic plaque lesions, identification of risk and susceptibility factors through the exploitation of longitudinal cohort data and multiomics and disintegration of carotid artery disease phenotypes into endotypes through joint modeling of multipleomics data sets and systems medicine approaches. Finally such stratification model will be validated and adjusted in the Taxinomisis clinical trial.

DETAILED DESCRIPTION:
Aim of the trial is to validate TAXINOMISIS system for risk stratification of carotid artery stenotic disease. Primary endpoints are stroke, transitory ischemic attack or retinal symptom while secondary endpoints are MRI silent brain lesions and carotid plaque progression.

Patient with moderate to severe extra-cranial, both asymptomatic and symptomatic, carotid artery stenosis will be enrolled in the prospective observational multi-center trial in five European (Athens, Barcelona, Belgrade, Genoa, Munich and Utrecht) vascular centers. Inclusion will last from 31.3.2018 - 01.06.2019. Patients with short life expectancy, high potential of stroke from other cause or patients with complex and tandem carotid lesions will be excluded from the trial.

Included patients will be examined clinically, basic laboratory exam will be performed and part of blood specimen will be stored and assessed later. Carotid plaque will be analysed by means of duplex and MRI image while brain lesions will be detected on brain MRI.

Treatment strategy will be dependent on guidelines of good clinical practice and let independently to institutional multidisciplinary panelist board. In patients treated with carotid endarterectomy (CEA) carotid plaque will be stored and assessed for future analysis. In respect to allocated therapy patients will follow different follow up protocols.

Intervention group: Patients undergoing intervention CEA or carotid artery stenting (CAS), will be followed by clinical examination and carotid duplex on 12, 24 and 36 month. If there is coexisting contralateral carotid stenosis greater than 50% and not requiring interventional treatment (CEA or CAS), patient should cross in optimal medical therapy group.

Optimal medical therapy group: Patients not subjected to intervention (or in whom one carotid has been treated with CAS or CEA and contra-lateral stenosis is greater than 50%) will be followed with carotid duplex (at 12, 24 and 36 months) and MRI imaging of carotid tree from aortic arch up to the circle of Willis after 12 and 36 months.

Trial plans to recruit 270 patients distributed in participating centers based on individual capabilities of each center. The diagnostic performance of the new risk model, and its accuracy to discriminate high versus low risk cases for cerebrovascular complications from carotid artery disease will be evaluated using Receiver Operating Characteristic (ROC) curve analysis. The accuracy (discriminated ability) of the model will be assessed by measuring the Area under the ROC curve (AUC). An AUC 0.80 and 90% CI, for the sensitivity of prediction model of 80% with marginal error of 10%, will be targeted.

Trial will terminate after finalizing 36 months of follow up for included patients at June 2022.

ELIGIBILITY:
Inclusion Criteria:

* Extracranial carotid stenosis greater than 50% stenosis (NASCET) in the carotid bifurcation or internal carotid artery assessed by means of ultrasound;
* Ability of the patient for follow-up examinations;
* Personally signed informed consent

Exclusion Criteria:

* Previous haemorrhagic stroke,
* Non-atherosclerotic carotid stenosis (e.g. dissection, floating thrombus, fibromuscular dysplasia, postirradiation lesion)
* Presence of stenotic lesions in the proximal common carotid artery,
* Recurrent carotid stenosis after CEA or CAS,
* Carotid aneurysm
* Bilateral carotid occlusion,
* Severe aortic arch calcifications and shaggy aorta
* Intracranial angioma or aneurysms,
* Severe pre-existing disability (modified Rankin scale ≥ 3);
* Contraindications for heparin, ASA and clopidogrel therapy
* Contraindication for MRI examination (metal implants, claustrophobia);
* Increased risk of thrombotic or embolic events (congenital or acquired thrombotic conditions, active untreated cancer, atrial fibrillation, severe cardiomyopathy with ejection fraction lower than 30%);
* Planned major surgery and/or life expectancy less than 3 years

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with extracranial carotid stenosis greater than 50% stenosis (NASCET) in the carotid bifurcation or internal carotid artery assessed by means of ultrasound
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Combined stroke, transitory ischemic attach and retinal transitory ischemic attach | 3 years
  rapidly developing clinical signs of focal (or global) disturbance of cerebral function, lasting more than 24 hours or leading to death, with no apparent cause other than that of vascular origin with CT or MRI confirmation of ischemia

SECONDARY OUTCOMES:
Silent brain lesions | 3 years
  ischemic lesions in the brain

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Fotiadis, PhD, Study Director — University of Ionania
Locations (4):
- University of Munich, Munich, Germany
- University of Utrecht, Utrecht, Netherlands
- Clinic for Vascular and Endovascular Surgery, Serbian Clinical Centre, Belgrade, Serbia, Serbia
- University of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided